CLINICAL TRIAL: NCT00036387
Title: A Randomized, Double-blind Trial of the Safety of Anti-TNF Chimeric Monoclonal Antibody (Infliximab) in Combination With Methotrexate Compared to Methotrexate Alone in Patients With Rheumatoid Arthritis on Standard Disease-modifying Anti-Rheumatic Drug Background Therapy.
Brief Title: A Study of the Safety and Effectiveness of Infliximab (Remicade) in Patients With Rheumatoid Arthritis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003133
Record Dates: First submitted 2002-05-09; First posted 2002-05-10 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-05

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid arthritis; infliximab; anti-TNF; methotrexate; safety and efficacy; Remicade
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab

INTERVENTIONS:
Drug: Infliximab

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of Infliximab (Remicade) in patients with Rheumatoid Arthritis. Infliximab (Remicade) targets specific proteins in the body's immune system to help control the development of inflammation to help reduce the pain of rheumatoid arthritis.

DETAILED DESCRIPTION:
This is a randomized (patients are assigned different treatments based on chance), double-blind (neither the patient nor the physician knows whether drug or placebo is being taken, or at what dosage) trial of the safety of anti-tumor necrosis factor (TNF) chimeric monoclonal antibody (Infliximab) in combination with methotrexate (MTX) compared to methotrexate alone in patients with rheumatoid arthritis on standard disease-modifying anti-rheumatic drug background therapy. The purpose of the study is to better understand the safety and occurrence of infections in patients treated with either placebo or 3 mg/kg and 10 mg/kg of infliximab in combination with methotrexate (MTX).

Patients will receive infusions of either placebo or 3 to 10mg/kg Infliximab at weeks 0, 2, 6, and 14 then every 8 weeks through week 46.

Safety evaluations will be performed at specified intervals throughout the study and will consist of laboratory tests, vital signs (such as blood pressure), physical examinations and the occurrence and severity of adverse events as well as other study specific procedures. Patients will receive 3 to10mg/kg Infliximab (Remicade) or placebo via infusion at weeks 0, 2, 6, and 14 then every 8 weeks through week 46.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of Rheumatoid Arthritis at least 3 months before screening
* If the patient is of childbearing potential, must have been using adequate birth control measures
* Patients must be receiving MTX for =3 months before randomization and at a stable dose(=25 mg/week) for =4 weeks before randomization

Exclusion Criteria:

* Patients must not be pregnant, nursing, or planning a pregnancy within 18 months of enrollment
* Patients must not have rheumatic disease other than Rheumatoid Arthritis or had any systemic inflammatory condition
* Patients must not be confined to a wheelchair
* Patients must not be treated with any approved or investigational biologic agent except for approved vaccines for immunizations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with serious infections occurring over the first 22 weeks of the trial

SECONDARY OUTCOMES:
The proportion of patients with infections & atypical/opportunistic infections. The duration of most frequently reported infections. Proportion of patients achieving ACR 20 criteria at 22 weeks. Effect of 1.5 mg/kg dose increment in reducing disease

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.

REFERENCES:
- [Result] Han C, Smolen JS, Kavanaugh A, van der Heijde D, Braun J, Westhovens R, Zhao N, Rahman MU, Baker D, Bala M. The impact of infliximab treatment on quality of life in patients with inflammatory rheumatic diseases. Arthritis Res Ther. 2007;9(5):R103. doi: 10.1186/ar2306. PMID 17922913
- [Result] Rahman MU, Strusberg I, Geusens P, Berman A, Yocum D, Baker D, Wagner C, Han J, Westhovens R. Double-blinded infliximab dose escalation in patients with rheumatoid arthritis. Ann Rheum Dis. 2007 Sep;66(9):1233-8. doi: 10.1136/ard.2006.065995. Epub 2007 Mar 28. PMID 17392352
- [Result] Westhovens R, Yocum D, Han J, Berman A, Strusberg I, Geusens P, Rahman MU; START Study Group. The safety of infliximab, combined with background treatments, among patients with rheumatoid arthritis and various comorbidities: a large, randomized, placebo-controlled trial. Arthritis Rheum. 2006 Apr;54(4):1075-86. doi: 10.1002/art.21734. PMID 16572442
- See also: A Study of the Safety and Effectiveness of Infliximab (Remicade) in Patients With Rheumatoid Arthritis. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=144&filename=CR003133_CSR.pdf